CLINICAL TRIAL: NCT02403557
Title: Individually-tailored Internet-delivered Cognitive Behaviour Therapy Treatment for Older Adults With Anxiety and Depression: a Randomized Controlled Trial
Brief Title: Internet-delivered Cognitive Behaviour Therapy for Older Adults With Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GA-Forte-Older-Adults-Anx
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Waiting Lists

ARMS (2):
- Tailored Internet-delivered CBT (Experimental): Tailored Internet-delivered CBT during 8 weeks.
  Interventions: Behavioral: Tailored Internet-delivered CBT
- Waitlist (Active Comparator): Weekly check-up.
  Interventions: Behavioral: Waitlist

INTERVENTIONS:
Behavioral: Waitlist — Weekly check up.
  Arms: Waitlist
Behavioral: Tailored Internet-delivered CBT — Tailored Internet-delivered CBT during 8 weeks.
  Arms: Tailored Internet-delivered CBT

SUMMARY:
The purpose of this study is to determine whether tailored internet-administrated cognitive behaviour therapy (ICBT) is a feasible approach in the treatment of anxiety symptoms and comorbid depressive symptoms in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Have anxiety symptoms

Exclusion Criteria:

* Suicidal ideation
* Alcohol addiction
* Other major primary psychiatric disorder
* Ongoing psychological treatment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Beck Anxiety Inventory (BAI) | Two weeks pre treatment, two weeks post treatment and 12 months post treatment
  Change from baseline in symptoms two weeks post treatment and at 12 months post treatment.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ) | Two weeks pre treatment, two weeks post treatment and 12 months post treatment
  Change from baseline in symptoms two weeks post treatment and at 12 months post treatment.
The Generalized Anxiety Disorder 7-item Scale (GAD-7) | Two weeks pre treatment, two weeks post treatment and 12 months post treatment
  Change from baseline in symptoms two weeks post treatment and at 12 months post treatment.
Quality of Life Inventory (QOLI) | Two weeks pre treatment, two weeks post treatment and 12 months post treatment
  Change from baseline in symptoms two weeks post treatment and at 12 months post treatment.
Montgomery Åsberg Depression Rating Scale - Self Rated (MADRS-S) | Two weeks pre treatment, two weeks post treatment and 12 months post treatment
  Change from baseline in symptoms two weeks post treatment and at 12 months post treatment.
Clinical Outcome in Routine Evaluation - Outcome Measure (CORE-OM) | Two weeks pre treatment, two weeks post treatment and 12 months post treatment
  Change from baseline in symptoms two weeks post treatment and at 12 months post treatment.
Cognitive Failures Questionnaire (CFQ) | Two weeks pre treatment, two weeks post treatment and 12 months post treatment
Wisconsin Card Sorting Test-64 (WCST-64) | Two weeks pre treatment, two weeks post treatment and 12 months post treatment